CLINICAL TRIAL: NCT00771680
Title: Evaluation of Effectiveness and Safety of Levemir® (Insulin Detemir), NovoMix® (Biphasic Insulin Aspart) and/or NovoRapid® (Insulin Aspart) in Insulin naïve Subjects With Type 2 Diabetes.
Brief Title: Observational Study to Evaluate the Effectiveness and Safety of Levemir®, NovoMix® 30 and NovoRapid® in Insulin naïve Subjects With Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: INS-3655
Record Dates: First submitted 2008-10-09; First posted 2008-10-13 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir; insulin aspart, insulin aspart protamine drug combination 30:70; Insulin Aspart

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: insulin detemir; Drug: biphasic insulin aspart 30; Drug: insulin aspart

INTERVENTIONS:
Drug: insulin detemir — Start dose and frequency at the discretion of the physician following clinical practice
Drug: biphasic insulin aspart 30 — Start dose and frequency at the discretion of the physician following clinical practice
Drug: insulin aspart — Start dose and frequency at the discretion of the physician following clinical practice

SUMMARY:
This study is conducted in Europe and Asia. The aim of this observational study is to evaluate the effectiveness and the incidence of serious adverse reactions while using Levemir®, NovoMix® and/or NovoRapid® in subjects with type 2 diabetes that have not used insulin previously under normal clinical practice conditions.

ELIGIBILITY:
Inclusion Criteria:

* Any insulin näive type 2 diabetic patient that able to use the drug as judged by the investigator

Exclusion Criteria:

* In accordance with approved label

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients of both genders who, in practice settings, have been deemed appropriate to receive Levemir®, NovoMix® 30 or and/or NovoRapid® as new treatment and as part of routine out-patient care by the prescribing physician.
Sampling Method: Non-Probability Sample
Enrollment: 10408 (Actual)
Dates: Start 2008-10; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
HbA1c | at baseline visit and during 3, 6, 9 and 12 months
Serious adverse drug reactions including major hypoglycaemic events | during 12 months of treatment

SECONDARY OUTCOMES:
Number of serious adverse drug reactions | during 12 months of treatment
Number of all major (daytime and nocturnal) hypoglycaemic events | during 12 months of treatment
Number of all minor (daytime and nocturnal) hypoglycaemic events | During 4 weeks prior to each study visit
Weight (BMI) change | At 6 and 12 months
Variability in fasting blood glucose values and average (mean) fasting blood glucose level | At baseline visit and after 6 and 12 months treatment
Average post-prandial blood glucose level (2h after dinner) | At baseline visit and after 6 and 12 months treatment
Quality of Life (QoL) as assessed by patient questionnaire | At baseline and the end of 6 and 12 months treatment

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (2):
- Novo Nordisk Investigational Site, Moscow, Russia
- Novo Nordisk Investigational Site, Kiev, Ukraine

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com